CLINICAL TRIAL: NCT02926482
Title: Test of a Workforce Development Intervention to Expand Buprenorphine Prescribers
Brief Title: Intervention to Expand Opioid Use Disorder Treatment Pharmacotherapy Prescribers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-0486; 1R01DA041415 (NIH); A195010 (Other: UW, Madison); ENGR/INDUSTRIAL ENGR (Other: UW, Madison)
Record Dates: First submitted 2016-09-09; First posted 2016-10-06 (Estimated); Last update posted 2024-08-13 (Actual); Status verified 2020-10

CONDITIONS: Opioid-use Disorder
Keywords: Evidence-based practice implementation; Buprenorphine; Addiction treatment; Extended-release naltrexone; Addiction
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): This arm will include 35 organizations who receive access to the Prescriber Recruitment Bundle (PRB) materials online via a secure website.
- PRB: organizations implementing the PRB (Experimental): This arm will include 35 organizations that will implement the intervention, the Prescriber Recruitment Bundle (PRB) using the NIATx Organizational Change Model (a model developed by our center research team).
  Interventions: Behavioral: Prescriber Recruitment Bundle (PRB)

INTERVENTIONS:
Behavioral: Prescriber Recruitment Bundle (PRB) — The Prescriber Recruitment Bundle (PRB) is a bundle pharmacotherapy capacity building practices. The PRB to be implemented contains the following elements, a) candidate identification strategies, b) prescriber education forums, c) prescriber-friendly workflow and risk-reduction strategies, d) academic detailing to recruit OUD prescribers, e) telemedicine, and f) organizational leadership and culture to support building OUD pharmacotherapy capacity.
  Other Names: PRB
  Arms: PRB: organizations implementing the PRB

SUMMARY:
This is a cluster-randomized controlled trial designed to increase the availability of buprenorphine and extended-release naltrexone treatment capacity for opioid use disorder (OUD). The intervention being tested is a bundle of OUD pharmacotherapy capacity building practices called the Prescriber Recruitment Bundle (PRB). For the study, 70 organizations will be identified and recruited, and those organizations will then be randomized into one of two arms: 1) control, and 2) intervention: organizations implementing the PRB using the Network for Improvement of Addiction Treatment (NIATx) Organizational Change Model. The primary research question is to test the impact of the PRB, relative to the control, on increasing buprenorphine treatment slots and extended-release naltrexone capacity and the number of patients receiving these pharmacotherapies.

DETAILED DESCRIPTION:
Overdoses due to non-medical use of prescription opioids and other opiates have become the leading cause of accidental deaths in the United States. Buprenorphine and extended-release naltrexone are key evidence-based interventions available to addiction treatment providers to treat opioid use disorder (OUD) and prevent overdose deaths. However, organizations' efforts to provide these pharmacotherapies have been hindered by limited success in recruiting providers (physicians, nurse practitioners, and physician assistants) to prescribe the medications. The addiction field has not historically attracted physicians and limits on access are compounded by buprenorphine's unique regulatory situation, in which physicians and other prescribers must apply for a waiver that allows them buprenorphine prescribing slots to treat 30 patients in the first year and 100 in the following years.

This study will address this emerging need to increase access to buprenorphine and extended-release naltrexone by testing a bundle of practices, called the Prescriber Recruitment Bundle (PRB), which aims to recruit prescribers licensed to prescribe buprenorphine to work with addiction treatment organizations. The PRB consists of the following elements, a) candidate identification strategies, b) prescriber education forums, c) prescriber-friendly workflow and risk-reduction strategies, d) academic detailing to recruit OUD prescribers, e) telemedicine to provide access to OUD pharmacotherapies, and f) organizational leadership and culture to support building OUD pharmacotherapy capacity.

In this cluster randomized controlled trial, the primary research question is to test the impact of the PRB implemented in conjunction with the NIATx organizational change model, relative to the control, on increasing the number of buprenorphine treatment slots and extended-release naltrexone capacity and increasing the number of patients receiving buprenorphine and extended-release naltrexone in the participating addiction treatment organizations. The secondary research question is to test if the PRB affects factors likely to be associated with prescriber recruitment, including: resources dedicated to prescriber recruitment, prescriber recruiter motivation, and current employed physician satisfaction. Lastly, qualitative methods will be used to study the context and processes that influence PRB adoption and fidelity and to understand and develop a deeper understanding of how the PRB influences recruitment beyond the existing study variables.

ELIGIBILITY:
Inclusion Criteria:

* Organizations that are publicly funded through the Substance Abuse and Prevention Treatment (SAPT) block grant, and had more than 100 admissions/annum about their interest in greater buprenorphine prescribing capacity.
* Organizations in the states of Florida, Ohio, and Wisconsin.

Exclusion Criteria:

* Organizations that are not publicly funded through the SAPT block grant, or do not have interest in expanding their buprenorphine prescribing capacity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Buprenorphine slots and extended naltrexone capacity survey | Monthly; beginning in Month 13 (April 2017) and continuing up to Month 50.
  Monthly number of assigned and open buprenorphine slots as well as extended-release naltrexone capacity and administrations over the past month.

SECONDARY OUTCOMES:
Organizational survey | Annual data collection, starting in Month 13 (April 2017) and continuing to Month 38.
  Measures PRB implementation fidelity
Physician Satisfaction | Annual data collection; starting in Month 13 (April 2017) and continuing up to Month 38.
  Collected via the "Physician Worklife Survey." Quantitative measure of a physician (or other prescribers) job satisfaction.
Qualitative surveys | Twice; first in Month 22 (January 2018) and again in Month 43.
  Measure of an addiction treatment organization's resources dedicated to prescriber recruitment. Participants will read statements regarding their organization's resources dedicated to prescriber recruitment, and their responses are recorded on a scale of 1-5, where 1 corresponds to "Not True" or "Strongly Disagree" and 5 corresponds to "Very True" or "Strongly Agree."

CONTACTS AND LOCATIONS:
Overall Officials: Todd Molfenter, Principal Investigator — Center for Health Enhancement Systems Studies, University of Wisconsin-Madison
Locations (3):
- United States (3):
  - Florida Alcohol and Drug Abuse Association, Tallahassee, Florida
  - Ohio Department of Mental Health and Addiction Services, Columbus, Ohio
  - Center for Health Enhancement Systems, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LH, Hedegaard H, Warner M. Drug-poisoning Deaths Involving Opioid Analgesics: United States, 1999-2011. NCHS Data Brief. 2014 Sep;(166):1-8. PMID 25228059
- [Background] Berglund M. A better widget? Three lessons for improving addiction treatment from a meta-analytical study. Addiction. 2005 Jun;100(6):742-50. doi: 10.1111/j.1360-0443.2005.01106.x. PMID 15918803
- [Background] Mattick RP, Breen C, Kimber J, Davoli M. Buprenorphine maintenance versus placebo or methadone maintenance for opioid dependence. Cochrane Database Syst Rev. 2014 Feb 6;2014(2):CD002207. doi: 10.1002/14651858.CD002207.pub4. PMID 24500948
- [Background] Jones CM, Campopiano M, Baldwin G, McCance-Katz E. National and State Treatment Need and Capacity for Opioid Agonist Medication-Assisted Treatment. Am J Public Health. 2015 Aug;105(8):e55-63. doi: 10.2105/AJPH.2015.302664. Epub 2015 Jun 11. PMID 26066931
- [Background] Molfenter T, Kim JS, Quanbeck A, Patel-Porter T, Starr S, McCarty D. Testing use of payers to facilitate evidence-based practice adoption: protocol for a cluster-randomized trial. Implement Sci. 2013 May 10;8:50. doi: 10.1186/1748-5908-8-50. PMID 23663749
- [Background] Molfenter T, Sherbeck C, Zehner M, Starr S. Buprenorphine Prescribing Availability in a Sample of Ohio Specialty Treatment Organizations. J Addict Behav Ther Rehabil. 2015;4(2):1000140. doi: 10.4172/2324-9005.1000140. PMID 26380328
- [Background] Stein BD, Gordon AJ, Dick AW, Burns RM, Pacula RL, Farmer CM, Leslie DL, Sorbero M. Supply of buprenorphine waivered physicians: the influence of state policies. J Subst Abuse Treat. 2015 Jan;48(1):104-11. doi: 10.1016/j.jsat.2014.07.010. Epub 2014 Aug 2. PMID 25218919
- [Background] Klein KJ, Conn AB, Sorra JS. Implementing computerized technology: an organizational analysis. J Appl Psychol. 2001 Oct;86(5):811-24. doi: 10.1037/0021-9010.86.5.811. PMID 11596799
- [Background] Tremblay MA, Blanchard CM, Taylor S, Pelletier LG, Villeneuve M. Work Extrinsic and Intrinsic Motivation Scale: Its value for organizational psychology research. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement. 2009;41(4):213-226.
- [Background] Williams ES, Konrad TR, Linzer M, McMurray J, Pathman DE, Gerrity M, Schwartz MD, Scheckler WE, Van Kirk J, Rhodes E, Douglas J. Refining the measurement of physician job satisfaction: results from the Physician Worklife Survey. SGIM Career Satisfaction Study Group. Society of General Internal Medicine. Med Care. 1999 Nov;37(11):1140-54. doi: 10.1097/00005650-199911000-00006. PMID 10549616
- [Background] Centers for Disease Control and Prevention (CDC). Vital Signs: Opioid painkiller prescribing. 2014.
- [Background] Soumerai SB, Avorn J. Principles of educational outreach ('academic detailing') to improve clinical decision making. JAMA. 1990 Jan 26;263(4):549-56. PMID 2104640
- [Background] Goldstein MG, Niaura R, Willey C, Kazura A, Rakowski W, DePue J, Park E. An academic detailing intervention to disseminate physician-delivered smoking cessation counseling: smoking cessation outcomes of the Physicians Counseling Smokers Project. Prev Med. 2003 Feb;36(2):185-96. doi: 10.1016/s0091-7435(02)00018-x. PMID 12590994
- [Background] McCarty D, Gustafson DH, Wisdom JP, Ford J, Choi D, Molfenter T, Capoccia V, Cotter F. The Network for the Improvement of Addiction Treatment (NIATx): enhancing access and retention. Drug Alcohol Depend. 2007 May 11;88(2-3):138-45. doi: 10.1016/j.drugalcdep.2006.10.009. Epub 2006 Nov 28. PMID 17129680
- [Background] Hoffman KA, Ford JH 2nd, Choi D, Gustafson DH, McCarty D. Replication and sustainability of improved access and retention within the Network for the Improvement of Addiction Treatment. Drug Alcohol Depend. 2008 Nov 1;98(1-2):63-9. doi: 10.1016/j.drugalcdep.2008.04.016. Epub 2008 Jun 18. PMID 18565693
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Raudenbush SW, Liu X. Statistical power and optimal design for multisite randomized trials. Psychol Methods. 2000 Jun;5(2):199-213. doi: 10.1037/1082-989x.5.2.199. PMID 10937329
- [Background] Knudsen HK, Abraham AJ, Roman PM. Adoption and implementation of medications in addiction treatment programs. J Addict Med. 2011 Mar;5(1):21-7. doi: 10.1097/ADM.0b013e3181d41ddb. PMID 21359109
- [Background] Singer JD, Willett JB. Applied longitudinal data analysis: modeling change and event occurrence. New York, NY: Oxford University Press; 2003.
- [Background] MacKinnon DP. Introduction to statistical mediation analysis. New York, NY: Lawrence Erlbaum Associates; 2008.
- [Background] Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. Psychol Methods. 2010 Dec;15(4):309-34. doi: 10.1037/a0020761. PMID 20954780
- [Background] Burke WW, Litwin GH. A causal model of organizational performance and change. In: Burke WW, Lake DG, Paine JW, eds. Organizational change: A comprehensive reader. San Francisco, CA: Jossey-Bass; 2009:273-299.
- [Background] Substance Abuse and Mental Health Services Administration, Center for Behavioral Health Statistics and Quality. Treatment Episode Data Set (TEDS): 2002-2012. National Admissions to Substance Abuse Treatment Services. Rockville, MD: Substance Abuse Mental Health Services Administration;2014.
- [Background] Fudala PJ, Bridge TP, Herbert S, Williford WO, Chiang CN, Jones K, Collins J, Raisch D, Casadonte P, Goldsmith RJ, Ling W, Malkerneker U, McNicholas L, Renner J, Stine S, Tusel D; Buprenorphine/Naloxone Collaborative Study Group. Office-based treatment of opiate addiction with a sublingual-tablet formulation of buprenorphine and naloxone. N Engl J Med. 2003 Sep 4;349(10):949-58. doi: 10.1056/NEJMoa022164. PMID 12954743
- [Background] Horgan CM, Reif S, Hodgkin D, Garnick DW, Merrick EL. Availability of addiction medications in private health plans. J Subst Abuse Treat. 2008 Mar;34(2):147-56. doi: 10.1016/j.jsat.2007.02.004. Epub 2007 May 17. PMID 17499959
- [Background] Schroeder SA. An agenda to combat substance abuse. Health Aff (Millwood). 2005 Jul-Aug;24(4):1005-13. doi: 10.1377/hlthaff.24.4.1005. PMID 16012140
- [Background] Alderks CE. Trends in the Use of Methadone and Buprenorphine at Substance Abuse Treatment Facilities: 2003 to 2011. 2013 Apr 23. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK384659/ PMID 27606405
- [Background] Knudsen HK, Abraham AJ, Oser CB. Barriers to the implementation of medication-assisted treatment for substance use disorders: the importance of funding policies and medical infrastructure. Eval Program Plann. 2011 Nov;34(4):375-81. doi: 10.1016/j.evalprogplan.2011.02.004. Epub 2011 Mar 2. PMID 21371752
- [Derived] Knudsen HK, Brown R, Jacobson N, Horst J, Kim JS, Kim H, Madden LM, Haram E, Molfenter T. Prescribers' satisfaction with delivering medications for opioid use disorder. Subst Abuse Treat Prev Policy. 2021 Oct 18;16(1):78. doi: 10.1186/s13011-021-00413-7. PMID 34663379
- [Derived] Knudsen HK, Brown R, Jacobson N, Horst J, Kim JS, Collier E, Starr S, Madden LM, Haram E, Toy A, Molfenter T. Physicians' satisfaction with providing buprenorphine treatment. Addict Sci Clin Pract. 2019 Aug 26;14(1):34. doi: 10.1186/s13722-019-0163-3. PMID 31446893
- [Derived] Molfenter T, Knudsen HK, Brown R, Jacobson N, Horst J, Van Etten M, Kim JS, Haram E, Collier E, Starr S, Toy A, Madden L. Test of a workforce development intervention to expand opioid use disorder treatment pharmacotherapy prescribers: protocol for a cluster randomized trial. Implement Sci. 2017 Nov 15;12(1):135. doi: 10.1186/s13012-017-0665-x. PMID 29141653